CLINICAL TRIAL: NCT00320099
Title: Phase 3 Study of Corticotherapy (Hydrocortisone Alone Versus Hydrocortisone Plus Fludrocortisone) Versus Corticotherapy Plus Intensive Insulin Therapy for Septic Shock
Brief Title: Combination of Corticotherapy and Intensive Insulin Therapy for Septic Shock
Acronym: COIITSS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Versailles (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Djillali Annane, AP-HP - University of Versailles SQY
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: AOM04100; P040421
Record Dates: First submitted 2006-04-27; First posted 2006-05-03 (Estimated); Last update posted 2010-04-06 (Estimated); Status verified 2010-04

CONDITIONS: Septic Shock
Keywords: septic shock; adrenal insufficiency; glucose control; mineralocorticoids
MeSH Terms: conditions — Shock, Septic; Adrenal Insufficiency | interventions — Hydrocortisone; Fludrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Hydrocortisone and convention glycemic control
  Interventions: Drug: hydrocortisone
- 2 (Experimental): Hydrocortisone and fludrocortisone and conventional glucose control
  Interventions: Drug: hydrocortisone; Drug: fludrocortisone
- 3 (Experimental): Hydrocortisone and intensive insulin therapy
  Interventions: Drug: recombinant human insulin; Drug: hydrocortisone
- 4 (Experimental): hydrocortisone, fludrocortisone and intensive insulin therapy
  Interventions: Drug: recombinant human insulin; Drug: hydrocortisone; Drug: fludrocortisone

INTERVENTIONS:
Drug: recombinant human insulin — intensive insulin therapy as a continuous infusion to maintain blood glucose levels between 4 and 6 mmol/l
  Arms: 3; 4
Drug: hydrocortisone — 50 mg as iv bolus every 6 hours for 7 days
Drug: fludrocortisone — 50 µg once a day via a nasogastric tube for seven days
  Arms: 2; 4
Drug: Hydrocortisone — hydrocortisone 50mg q6 for 7 days
  Arms: 1

SUMMARY:
This study will compare, in adults with septic shock, the safety and efficacy of a combination of moderate doses of corticosteroids and intensive insulin therapy to that of moderate doses of corticosteroids. In addition, this study will compare the efficacy and safety of hydrocortisone alone versus hydrocortisone plus fludrocortisone

DETAILED DESCRIPTION:
Objectives:

Comparison, in patients with septic shock, of efficacy and safety of the combination of moderate doses of corticosteroids and intensive insulin therapy to that of moderate doses of corticosteroids; and of efficacy and safety of hydrocortisone alone versus hydrocortisone plus fludrocortisone Methods

Study design :

This is a multicenter, prospective, randomised trial on parallel groups

Study treatments :

Experimental arm A:

A1=50 mg iv every 6 hours of hydrocortisone (hemisuccinate), 50µg through the nasogastric tube of 9 alpha fludrocortisone, for 7 days AND strict control of blood glucose levels with a target of 4,4 to 6 mmol/L using continuous iv infusion of insulin up to intensive care unit discharge.

A2=50 mg iv every 6 hours of hydrocortisone (hemisuccinate) for 7 days AND strict control of blood glucose levels with a target of 4,4 to 6 mmol/L using continuous iv infusion of insulin up to intensive care unit discharge.

Control arm B:

B1:50 mg iv every 6 hours of hydrocortisone (hemisuccinate), 50µg through the nasogastric tube of 9 alpha fludrocortisone, for 7 days.

B2:50 mg iv every 6 hours of hydrocortisone (hemisuccinate)for 7 days. Study Primary outcome : In-hospital mortality

Sample size calculation :

The expected in-hospital mortality rate in the control group is 50%. To detect an absolute reduction in in-hospital mortality rate of 12.5 %, that is 37.5% in the experimental arm versus 50% in the control arm, and considering risk alpha of 0,05 and a risk beta of 0,20, 254 patients per treatment arms are needed, for a total of 508 patients.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted in intensive care units for septic shock and meeting all following criteria

* Proven infection
* Need for vasopressor to maintain systemic arterial tension above 90 mmHg
* Multiple organ dysfunction as defined by a SOFA score ³ 8.
* Need for treatment with moderate dose of corticosteroids

Exclusion Criteria:

One of the following :

* Pregnancy
* Less than 18 years old
* Moribund (i.e. expected to die on day of intensive care unit admission)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | Day 180

SECONDARY OUTCOMES:
Secondary outcomes : | Day 180
90-day and 180-day mortality. | Day 180
Duration of life-supporting treatments (i.e. vasopressors and mechanical ventilation) | Day 180
Time to resolve multiple organ dysfunction, i.e. to obtain a SOFA score < 8 | Day 180
Hospital length of stay. | Day 180
Number of hypoglycaemic events (blood glucose < 4 mmol/l) during insulin infusion | Day 180
Muscle weakness at discharge from intensive care unit, 90-day and 180-day | Day 180
Post traumatic stress disorders | Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Djillali annane, MD, PhD, Study Chair — Assistance Publique Hôpitaux de Paris - University of Versailles
Locations (8):
- France (8):
  - Hôpital Avicenne, Bobigny
  - Hôpital Jean Verdier, Bondy
  - CHU Grenoble, Grenoble
  - Hôpital central, Nancy
  - Hôpital Saint Louis, Paris
  - Hôpital Bichat Claude Bernard, Paris
  - hôpital Cochin, Paris
  - Hôpital Delafontaine, Saint-Denis

REFERENCES:
- [Result] COIITSS Study Investigators; Annane D, Cariou A, Maxime V, Azoulay E, D'honneur G, Timsit JF, Cohen Y, Wolf M, Fartoukh M, Adrie C, Santre C, Bollaert PE, Mathonet A, Amathieu R, Tabah A, Clec'h C, Mayaux J, Lejeune J, Chevret S. Corticosteroid treatment and intensive insulin therapy for septic shock in adults: a randomized controlled trial. JAMA. 2010 Jan 27;303(4):341-8. doi: 10.1001/jama.2010.2. PMID 20103758